CLINICAL TRIAL: NCT02847065
Title: Study Single-center, Uncontrolled, Retrospective, the Association Between Advancing Age and Mortality at 30 Days in Patients With Bacteremia E. Coli Beta-lactamase Phenotype Extended Spectrum
Brief Title: The Association Between Advancing Age and Mortality at 30 Days in Patients With Bacteremia E. Coli Beta-lactamase Phenotype Extended Spectrum RC15_0421
Acronym: MoBaCo
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0421
Record Dates: First submitted 2016-07-21; First posted 2016-07-27 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Beta-lactamase Extended Spectrum, E. Coli, Elderly, Mortality, Risk Factor
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
In the US and Europe, bacteremia are ranked the 7th leading cause of death from all causes. E. coli is one of the main microorganism involved, responsible for 30% to 45% of bacteremia. In Europe, bacteremia E. coli, including BLSE phenotype, have a strong impact on public health, causing increased mortality, particularly in the elderly, and an increase in the average hospital stay. However, few studies have specifically concerned with the criteria associated with mortality of elderly patients with BLSE E. coli bacteremia. Finally, improving epidemiological knowledge of the elderly patients with bacteremia due to BLSE E. coli has importance in terms of public health and is a prerequisite to the development of preventive strategies and to improve the short-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* All patients with positive blood culture E. coli BLSE will be included in the study. Bacteremia E. coli BLSE will be defined as the identification of one or more blood cultures positive for E. coli BLSE in patients with clinical criteria of systemic inflammatory response, at least two of the following 4 criteria:

  * temperature> 38 ° C or < 36 ° C;
  * heart rate> 90 beat / min;
  * respiratory rate > 20 c / min or PaCO2 < 32 mmHg;
  * WBC > 12,000 / microL or < 4000 / microL or 10% immature forms

Exclusion Criteria:

* For each patient included, only the first episode of bacteremia will be included in the study

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All data concerning blood cultures analyzed in the bacteriology department of University Hospital of Nantes are stored digitally, particularly E. coli ESBL. Thus, the extraction of these data will allow the retrospective inclusion of patients and enhance the feasibility of the study.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Association between advancing age and mortality at 30 days in patients with bacteremia E. coli beta-lactamase phenotype extended spectrum. | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France